CLINICAL TRIAL: NCT05230147
Title: Hemodynamic Effects of Transcutaneous Spinal Cord Stimulation During Passive Orthostasis: a Prospective Single-center Randomized Cross-over Study
Brief Title: Spinal Cord Stimulation for Orthostatic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Ortho-stim_2022
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Orthostatic Hypotension
Keywords: spinal cord stimulation; hypotension; hemodynamic effects
MeSH Terms: conditions — Hypotension, Orthostatic; Hypotension | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will undergo spinal cord stimulation or a sham procedure during tilt testing following randomization. Then a second test will be performed the same day after crossover.
  A repeated test will be performed after 7 days in reverse order (sham or stimulation).
Who Masked: Investigator
Masking Description: Stimulation patches will be applied in all patients and simulating of stimulation will be provided by an audible order by an investigator. Since high-frequency stimulation is almost non-sensible, masking is possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal cord stimulation (Experimental): Before tilt testing, adhesive patches are applied to subjects' back skin. Single stimuli are delivered to the patches in order to define the stimulation threshold under the guidance of neuromyography. An investigator says loudly: "I am initiating high-frequency stimulation". Stimulation is initiated within 2 min before tilting the table. Then verticalization of the table 45 degrees is performed, and the test is continued for 15-30 min. Beat-to-beat blood pressure recording is carried out and 10 min after blood pressure complete stabilization the test is ended.
  Interventions: Procedure: Spinal cord stimulation
- Sham stimulation (Sham Comparator): Before tilt testing, adhesive patches are applied to subjects' back skin. Single stimuli are delivered to the patches in order to define stimulation threshold under the guidance of neuromyography. An investigator says loudly: "I am initiating high-frequency stimulation". No stimulation is initiated. Two minutes after, verticalization of the table 45 degrees is performed, and the test is continued for 15-30 min. Beat-to-beat blood pressure recording is carried out and 10 min after blood pressure complete stabilization the test is ended.
  Interventions: Procedure: Sham stimulation

INTERVENTIONS:
Procedure: Spinal cord stimulation — Single stimuli are delivered to define the stimulation threshold. High-frequency stimulation with modulated current via skin patches captures posterior horns of the spinal cord.
  Arms: Spinal cord stimulation
Procedure: Sham stimulation — Single stimuli are delivered to define the stimulation threshold. High-frequency stimulation is not delivered.
  Arms: Sham stimulation

SUMMARY:
This is a prospective single-center randomized crossover control study that aims to evaluate the effects of non-invasive transcutaneous spinal cord stimulation in patients with known or suspected orthostatic hypotension.

DETAILED DESCRIPTION:
The hypothesis is that transcutaneous spinal cord stimulation at thoracic level may correct hypotensive episodes during tilt testing in subjects with blood pressure drops.

Eligible patients will sign an informed consent form before the procedure. Non-invasive transcutaneous electrical stimulation of the spinal cord will be applied using modulated electrical impulses through external adhesive electrode patches connected to a neural stimulator device. The study protocol includes analysis of the following parameters: heart rate; 12-lead electrocardiogram; continuous beat-to-beat blood pressure recordings (measured noninvasively by plethysmography) before stimulation, during stimulation and after spinal cord stimulation. All registered data will be analyzed at the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years
2. Suspected orthostatic hypotension (having a history of syncope and/or pre-syncope that occurred during the transition to an upright position, with complaints of recurrent dizziness that occurs during the transition to an upright position) or documented orthostatic hypotension.
3. The patient who signed the informed consent form

Exclusion Criteria:

1. Orthostatic hypotension caused by acute hypovolemia or bleeding.
2. Chronic heart failure III-IV functional class (NYHA)
3. Structural heart disease of the following: hypertrophic cardiomyopathy with obstruction of the left ventricular outflow tract, acute coronary syndrome, restrictive cardiomyopathy, hemodynamically significant valvular heart defects, uncorrected hemodynamically significant congenital heart defects.
4. Ongoing acute illness.
5. >90% paced cardiac rhythm.
6. Permanent atrial fibrillation.
7. A history of transient ischemic attack or stroke within 3 months before the enrollment and/or incomplete recovery.
8. Pulmonary embolism <1 month ago.
9. Epilepsy.
10. The presence of an implantable pump.
11. Patients with contraindications to the use of the patch electrodes used in this study, as indicated in the relevant instructions for use.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure drop correction | 5-30 minutes following verticalization
  It is suggested that spinal cord stimulation will correct systolic blood pressure drop during tilt testing. The effect is expected within 5-10 mmHg as a difference between minimum systolic blood pressure during stimulation and without stimulation (sham).

SECONDARY OUTCOMES:
Diastolic blood pressure drop correction | 5-30 minutes following verticalization
  It is suggested that spinal cord stimulation will correct diastolic blood pressure drop during tilt testing. The effect is expected within 5-10 mmHg as a difference between minimum diastolic blood pressure during stimulation and without stimulation (sham).

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny N Mikhaylov, Assoc.prof., Principal Investigator — Almazov National Medical Research Centre; Evgeny V Shlyakhto, Prof, Study Chair — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed during regular meetings of the study and supervising committees after enrollment of at least 30% of subjects.

REFERENCES:
- [Background] Mikhaylov EN, Moshonkina TR, Zharova EN, Garkina SV, Kovzelev PD, Belyaeva NN, Kozlenok AV, Lebedev DS, Shlyakhto EV. Acute Cardiovascular Effects of Non-Invasive Electrical Spinal Cord Stimulation: Results from a Pilot Study in Humans. J Cardiovasc Transl Res. 2020 Dec;13(6):891-893. doi: 10.1007/s12265-020-10014-7. Epub 2020 May 6. PMID 32378161
- [Background] Lobov GI, Gerasimenko YP, Moshonkina TR. Mechanisms of Blood Flow Regulation in the Skin during Stimulation of the Spinal Cord in Humans. Dokl Biol Sci. 2019 Mar;485(1):27-29. doi: 10.1134/S0012496619020030. Epub 2019 Jun 13. PMID 31197588
- [Background] Phillips AA, Squair JW, Sayenko DG, Edgerton VR, Gerasimenko Y, Krassioukov AV. An Autonomic Neuroprosthesis: Noninvasive Electrical Spinal Cord Stimulation Restores Autonomic Cardiovascular Function in Individuals with Spinal Cord Injury. J Neurotrauma. 2018 Feb 1;35(3):446-451. doi: 10.1089/neu.2017.5082. Epub 2017 Nov 21. PMID 28967294